CLINICAL TRIAL: NCT06381102
Title: How Does the Length of Pulse Trains and Pulse Intervals Affect Tolerability With Transcutaneous Auricular Vagus Nerve Stimulation?
Brief Title: Transcutaneous Vagus Nerve Stimulation (taVNS) Dosage Study 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Marlon Wong, Associate Professor of Clinical, University of Miami
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 20240134
Record Dates: First submitted 2024-04-19; First posted 2024-04-24 (Actual); Results first posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- taVNS 30/30 group (Experimental): Participants in the group taVNS 30/30 will be in this group for up to 3 hours.
  Interventions: Device: transcutaneous auricular vagus nerve stimulation 30/30
- taVNS 10/10 group (Experimental): Participants in the group taVNS 10/10 will be in this group for up to 3 hours.
  Interventions: Device: transcutaneous auricular vagus nerve stimulation 10/10

INTERVENTIONS:
Device: transcutaneous auricular vagus nerve stimulation 30/30 — Transauricular vagus nerve stimulation (taVNS) is a simple technique in which small surface electrodes are placed over the skin of the ear that are thought to be innervated by the auricular branch of the vagus nerve (ABVN). Participants in this group will first receive taVNS with a 30 second on and 30 second off, for 1 hour, in-person.
  Arms: taVNS 30/30 group
Device: transcutaneous auricular vagus nerve stimulation 10/10 — Transauricular vagus nerve stimulation (taVNS) is a simple technique in which small surface electrodes are placed over the skin of the ear that are thought to be innervated by the auricular branch of the vagus nerve (ABVN). Participants in this group will first receive taVNS with a 10 second on and 10 second off, for 1 hour, in-person.
  Arms: taVNS 10/10 group

SUMMARY:
The purpose of this research study is to investigate the effects of different forms of a gentle form of electrical stimulation applied to the ear, known as transcutaneous auricular vagus nerve stimulation (taVNS). The research team is interested in how the different forms affect comfort and tolerability, as well as how well it works.

ELIGIBILITY:
Inclusion Criteria:

1. between the ages of 18-80 years
2. English speaking (must be able to consent and complete the interviews in English)

Exclusion Criteria:

1. chronic pain (average intensity >2/10 on 0-10 scale, for longer than 3 months)
2. acute pain of intensity greater than 3/10
3. chronic inflammatory conditions that are poorly controlled (e.g., diabetes, autoimmune disease)
4. any unstable medical condition or medical contraindication to moderate physical exertion (e.g., unstable angina or cardiac arrythmia)
5. pregnancy
6. currently taking Buprenorphine or recently stopped taking (within 1 month)
7. presence of cognitive impairment or language barrier that impairs full autonomy in the consent process or in the ability to participate in detailed interviews
8. implants in the head or neck, cochlear implants, or pacemaker
9. head or neck metastasis or recent ear trauma
10. history of epilepsy
11. history of autonomic nervous system dysfunction (e.g., postural orthostatic tachycardia syndrome).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2024-04-13 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marlon Wong, DPT, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants will be randomized in Period 1 to receive either taVNS 30/30 first or taVNS 10/10 first then the participants will washout for 5 days and will then switch and crossover in Period 2 to receive the opposite treatment from what they received in Period 1 which will be either the taVNS 30/30 first or the taVNS 10/10 first depending on what they were first originally randomized to in Period 1.
Period: Intervention 1
Arm/Group | taVNS 30/30 Group | taVNS 10/10 Group
Started | 17 | 14
Completed | 17 | 14
Not Completed | 0 | 0
Period: Washout 5 Days
Arm/Group | taVNS 30/30 Group | taVNS 10/10 Group
Started | 17 | 14
Completed | 17 | 12
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2
Period: Intervention 2
Arm/Group | taVNS 30/30 Group | taVNS 10/10 Group
Started | 17 | 12
Completed | 17 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | taVNS 30/30 Group | taVNS 10/10 Group | Total
Number analyzed (Participants) | 17 | 14 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.0 (13.0) | 29.2 (6.8) | 30.2 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 16
  Male | 8 | 7 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 7 | 11
  Not Hispanic or Latino | 13 | 7 | 20
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 13 | 12 | 25
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Tolerability Measured by Tolerability Questionnaire
Description: Tolerability will be assessed with a questionnaire with scores ranging from 0 -10 (with 0 being no irritation or discomfort and 10 being the worst possible irritation or discomfort) for irritation from tingling/tickling/pricking during taVNS.
Time Frame: 3 hours
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | taVNS 30/30 Group | taVNS 10/10 Group
Number analyzed (Participants) | 29 | 29
score on a scale | 2.2 (1.8) | 2.2 (1.8)

2. Primary Outcome: Tolerability Measured by Self-report
Description: The number of participants who reported mild pain with the intervention.
Time Frame: 3 hours
Measure: Count of Participants; unit: Participants
Arm/Group | taVNS 30/30 Group | taVNS 10/10 Group
Number analyzed (Participants) | 29 | 29
Participants | 7 | 8

3. Secondary Outcome: Change in Heart Rate Variability (HRV)
Description: HRV will be measured with an H10 chest strap device. Values after stimulation will be subtracted from baseline values; thus, a positive number will indicate an increase in HRV post taVNS measured in milliseconds.
Time Frame: Baseline and 3 hours
Measure: Mean (Standard Deviation); unit: Milliseconds
Groups:
- taVNS 30/30 Group: Participants in the group taVNS 30/30will be in this group for up to 3 hours.
  transcutaneous auricular vagus nerve stimulation 30/30: Transauricular vagus nerve stimulation (taVNS) is a simple technique in which small surface electrodes are placed over the skin of the ear that are thought to be innervated by the auricular branch of the vagus nerve (ABVN). Participants in this group will first receive taVNS with a 30 second on and 30 second off, for 1 hour, in-person.
Arm/Group | taVNS 30/30 Group | taVNS 10/10 Group
Number analyzed (Participants) | 29 | 29
Milliseconds | 7.2 (12.2) | 4.4 (12.1)

ADVERSE EVENTS:
Time Frame: 72 hours
Arm/Group | taVNS 30/30 Group | taVNS 10/10 Group
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/31
Other Adverse Events (participants affected / at risk) | 0/29 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-29): https://cdn.clinicaltrials.gov/large-docs/02/NCT06381102/Prot_SAP_000.pdf